CLINICAL TRIAL: NCT04637412
Title: Perceived Effectiveness of Added Sugar Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Center for Science in the Public Interest (CSPI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1641776
Record Dates: First submitted 2020-11-16; First posted 2020-11-19 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Health Knowledge; Attitude to Health
Keywords: Added Sugars; Health messaging

STUDY DESIGN:
Intervention Model Description: The study uses both a between- and within-subjects design.
  Between-subjects design: Participants will be randomized to view restaurant menu items with a control label (QR code) or either one of two added sugars labels: an icon based label or the same icon plus text. (Within the icon condition, participants will be randomized to view 1 of 6 label icons. In the icon plus text condition, participants will be randomized to see 1 of 3 text options accompanying 1 of the 6 icons.
  Within-subjects design:
  To identify which label is perceived as most discouraging, participants will view the 3 labels one-by-one in random order, for a total of 3 conditions.
  To identify which design variations in icon and text are perceived as most discouraging, participants will view 6 icon-only labels one-by-one in random order. Then participants will view each of the 3 text variations together with one of the icons one-by-one in random order.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control label (Experimental): Participant will see a QR code and footnote saying, "Scan the QR code for more menu information." The label will be applied to all menu items displayed.
  Interventions: Other: Menu label
- Icon plus text added sugars label (Experimental): Participant will see a label containing an icon plus text label with an explanatory footnote. The label will be applied to items high in added sugars (exceeding half the daily value). Participants will randomly view one of 18 variations of icons and text in this arm.
  Interventions: Other: Menu label
- Icon only added sugars label (Experimental): Participant will see a label containing an icon only with an explanatory footnote. The label will be applied to items high in added sugars (exceeding half the daily value). Participants will randomly view one of 6 variations of icons in this arm.
  Interventions: Other: Menu label

INTERVENTIONS:
Other: Menu label — Participants will be shown a sample of items from a restaurant menu, displayed with labels

SUMMARY:
This study aims to develop a restaurant menu label to indicate foods and beverage items on restaurant menus that contain high amounts of added sugars and to test its perceived effectiveness.

DETAILED DESCRIPTION:
Objectives and hypotheses:

The goal of this study is to examine how added sugar restaurant menu labels influence U.S. adults' perceptions and reactions. Predictions:

In a between-subjects experiment with 3 arms (control label, icon-only added sugars label, and icon plus text added sugars label):

1. Added sugar labels will be perceived as more effective than the control label.
2. The text plus icon label will be perceived as more effective than the icon-only label.
3. A larger proportion of participants who see the added sugar labels will report learning something new than those who see the control label.
4. Added sugar labels will lead participants to more accurately identify restaurant menu items high in added sugars compared to the control label, and the text plus icon label will outperform the icon-only label on this outcome.

Additionally, using a within-subjects design:

The study will examine which label (control, icon, text plus icon) most discourages wanting to consume menu items high in added sugars.

Analyses will compare various icon and text options for the added sugars label to determine which icon and which text variations are perceived as most discouraging for wanting to consume items high in added sugars. The is no hypothesis about which will be perceived as more discouraging.

Planned analyses:

For predictions 1-2: linear regression model (OLS) regressing PME on indicator variables for experimental condition. The margins command in STATA will be used to conduct pairwise comparisons between each condition (i.e., icon-only vs. icon plus text label). Also, PME will be regressed on an indicator variable combining the added sugar label groups.

For predictions 3-4, Poisson regression with robust standard errors will be used to estimate relative probability, regressing each dichotomous outcome on indicator variables for experimental condition. The margins command in STATA will be used to conduct pairwise comparisons between each condition. The outcomes will be regressed on an indicator variable combining the added sugar label groups. If the Poisson regressions do not converge, logistic regression will be used.

For the within-subjects comparisons, mixed effects linear models will be used to assess the relationship between condition and rating of label discouragement for consuming items high in added sugars.

A critical alpha 0.05 will be used, and statistical tests will be two-tailed. Because this is an initial, exploratory study to help identify the best performing label to use in a larger trial, alpha level will not be adjusted to control for multiple comparisons.

If there is evidence of deviations from modeling assumptions required for the parametric tests above, non-parametric sensitivity analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Equal or greater than 18 years of age
* Less than 100 years of age
* English-speaking
* U.S. residents
* Had to have purchased food from a restaurant at least once per month prior to the COVID-19 pandemic
* Participants will reflect the U.S. Census Bureau's 2018 American Community Survey 5-year estimates for gender, race/ethnicity, educational attainment, and age

Exclusion criteria:

* Failing the attention check question
* Completing the survey in less than 30% of the median completion time
* Straightlining
* Providing nonsensical responses to open-ended questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1448 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
Perceived message effectiveness (PME) | Up to approximately 5 minutes
  Measured using 3 items adapted from Baig et al. (2018): scale 1-5, "This label makes me concerned about the health effects of consuming menu items high in added sugars", "This label makes consuming menu items high in added sugars seem unpleasant", "This label discourages me from wanting to consume menu items high in added sugars." This outcome is for the between-subjects experiment.
Perception of how discouraging the label is for wanting to consume items high in added sugars | Up to approximately 7 minutes
  Based on a single item adapted from Baig et al. (2018): "This label discourages me from wanting to consume menu items high in added sugar" (scale 1-5). This outcome is the within-subjects objectives.
Perception of knowledge gain | Up to approximately 1 minute
  Dichotomous response (yes/no) to the question, "Did you learn something new from this label?" This outcome is for the between-subjects experiment.
Correct identification of items high in added sugars | Up to approximately 2 minutes
  "Now please look at the menu items below, and select all the ones you think have more than half the daily value for added sugars" with 8 possible responses. A dichotomous outcome variable based on the distribution of correct answers in the sample will be created. This outcome is for the between-subjects experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Falbe, ScD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baig SA, Noar SM, Gottfredson NC, Boynton MH, Ribisl KM, Brewer NT. UNC Perceived Message Effectiveness: Validation of a Brief Scale. Ann Behav Med. 2019 Jul 17;53(8):732-742. doi: 10.1093/abm/kay080. PMID 30321252
- [Derived] Sigala DM, Hall MG, Musicus AA, Roberto CA, Solar SE, Fan S, Sorscher S, Nara D, Falbe J. Perceived effectiveness of added-sugar warning label designs for U.S. restaurant menus: An online randomized controlled trial. Prev Med. 2022 Jul;160:107090. doi: 10.1016/j.ypmed.2022.107090. Epub 2022 May 17. PMID 35594928